CLINICAL TRIAL: NCT01946451
Title: Gene Expression and Their Correlations in Patients With Idiopathic and Secondary Epiretinal Membranes in Proliferative Diabetic Retinopathy
Brief Title: Gene Expression in Patients With Epiretinal Membranes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Dorota Romaniuk, MD, Medical University of Silesia
Other Study IDs: SilesianMU
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: idiopathic epiretinal membranes; secondary epiretinal membranes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Idiophatic ERMs
- Secondary ERMs

SUMMARY:
The purpose of this study was to investigate the expression of selected genes both in epiretinal membranes (ERMs) and peripheral blood mononuclear cells (PBMCs) from patients with primary and secondary epiretinal membranes in proliferative diabetic retinopathy. Possible correlations between messenger ribonucleic acid (mRNA) levels of these genes were also identified.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian race,
* both males and females,
* aged ≥ 55 years,
* suffering from idiopathic ERMs or secondary ERMs in proliferative diabetic retinopathy (PDR).
* Presence of ERM was proven in optical coherence tomography (OCT) examination.

Exclusion criteria:

* aged < 55 years,
* systemic connective tissue disease,
* active inflammatory process

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population description:
  The blood and ERM samples were obtained from patients treated in the Department of Ophthalmology, University Hospital No. 5, Medical University of Silesia, Katowice, Poland.
  All subjects underwent a complete ophthalmic examination: best corrected visual acuity (BCVA), tonometry, slit lamp examination of anterior and posterior segment, optical coherence tomography (OCT) of the central retina.
Sampling Method: Non-Probability Sample
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Gene expression in patients with idiopathic and secondary epiretinal membranes in proliferative diabetic retinopathy. | The period between the diagnosis of the ERMs and the actual surgery for the condition was between 2 and 43 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Silesia, Katowice, Poland